CLINICAL TRIAL: NCT06121206
Title: Altitude-like Cognition Training to Target Brain Erythropoietin as a Novel Mechanism of Long-lasting Neuroplasticity and Cognitive Functions
Brief Title: Effects of Altitude-like Cognition Training on Neuroplasticity and Cognitive Functions
Acronym: ALTIBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: European Research Council (Other); University of Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kamilla Woznica Miskowiak, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-22028111; P-2022-354 (Registry Identifier: Danish Data Protection Agency)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment; Bipolar Disorder; Depression
Keywords: Cognition; Neuroplasticity; Hypoxia; Cognitive training; Depression; Bipolar Disorder; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Bipolar Disorder; Depression; Hypoxia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Substudy 1: The study has a double-blinded design. Neither the participant nor the outcome assessors will know whether the participant is receiving (1) altitude-like hypoxia (12%) combined with cognitive training, (2) hypoxia with no training, (3) cognitive training under normoxia (20%), or (4) normoxia with no training.
  Substudy 2: The study has an assessor-blinded design. The outcome assessor will not know whether the participant is receiving (1) altitude-like hypoxia (12%) combined with cognitive training or (2) treatment as usual (TAU).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Altitude-like hypoxia (12%) combined with cognitive training (Experimental): Participants breathe 12% ambient oxygen in an altitude-training room, 3.5 hours daily, 5-6 days per week for 3 weeks. On iPads, they perform cognitive training, which is interleaved by short breaks.
  Interventions: Other: Altitude-like hypoxia (12% O2); Behavioral: Cognitive training
- Altitude-like hypoxia (12%) with no training (Active Comparator): Participants breathe 12% ambient oxygen in an altitude-training room, 3.5 hours daily, 6 days per week for 3 weeks. On iPads, they perform matched control games without cognitive benefits, which is interleaved by short breaks.
  Interventions: Other: Altitude-like hypoxia (12% O2); Behavioral: Sham training
- Normoxia (20%) combined with cognitive training (Active Comparator): Participants breathe 20% ambient oxygen in an altitude-training room, 3.5 hours daily, 6 days per week for 3 weeks. On iPads, they perform cognitive training, which is interleaved by short breaks.
  Interventions: Other: Normoxia (20% O2); Behavioral: Cognitive training
- Normoxia (20%) combined with no training (Sham Comparator): Participants breathe 20% ambient oxygen in an altitude-training room, 3.5 hours daily, 6 days per week for 3 weeks. On iPads, they perform matched control games without cognitive benefits, which is interleaved by short breaks.
  Interventions: Other: Normoxia (20% O2); Behavioral: Sham training
- Treatment as usual (No Intervention): Participants receive no additional care or intervention between baseline and end-of-treatment assessment points.

INTERVENTIONS:
Other: Altitude-like hypoxia (12% O2) — Fresh air with 12% O2, is blown into a sealed 20 m³ room by a 4kW air compressor with a safety-approved system developed by HöhenBalance, Austria. After participants enter the room, the O2 levels will be reduced from 16% to 12% (≈ 4,400 meters altitude) in a 30 minutes lead-in phase. The target O2 level of 12% will be maintained over three hours
  Arms: Altitude-like hypoxia (12%) combined with cognitive training; Altitude-like hypoxia (12%) with no training
Other: Normoxia (20% O2) — Fresh air with 20% O2, is blown into a sealed 20 m³ room by a 4kW air compressor with a safety-approved system developed by HöhenBalance, Austria. The target O2 level of 20% will be maintained over 3.5 hours
  Arms: Normoxia (20%) combined with cognitive training; Normoxia (20%) combined with no training
Behavioral: Cognitive training — The web-based cognitive training (Happy Neuron Pro) is grounded on principles of neuroplasticity-based learning by being intensive, neuroadaptive, engaging and rewarding. The active training involves parametric task adjustment by decreasing stimuli presentation time, increasing working memory load, decreasing time to respond, and increasing the number of non-target items (distractors).
  Arms: Altitude-like hypoxia (12%) combined with cognitive training; Normoxia (20%) combined with cognitive training
Behavioral: Sham training — Participants in the no training control condition receive computer games similar to Happy Neuron Pro but with low cognitive demand that produce no cognitive benefits. Specifically, this sham procedure involves the exact same stimuli as the active condition but with changes from trial to trial only in the appearance of the tasks.
  Arms: Altitude-like hypoxia (12%) with no training; Normoxia (20%) combined with no training

SUMMARY:
The goal of this clinical trial is to investigate the effects of a three-week altitude-like cognition training intervention in healthy individuals (substudy 1) and symptomatically stable patients with mood disorders (depression or bipolar disorder; substudy 2). This multi-modal intervention consists of an adaptive cognitive training programme that participants complete while they're inside an altitude-training room with 12% O2, corresponding to 4400 meters altitude.

Across substudy 1 and 2, the investigators hypothesize that altitude-like cognition training has a beneficial effect on cognition after three-weeks treatment completion measured with a global cognition composite score (primary outcome measure). Further, the investigators hypothesize that hypoxia and cognition training will yield improved executive functioning after treatment completion and changes in brain activity during working memory in the dorsal prefrontal cortex 4 weeks after treatment completion (secondary outcome measures). In the patient study, the investigators further hypothesize that the intervention will have beneficial effects on daily-life cognition measured in virtual reality (VR) 4 weeks after treatment completion (secondary outcome measure in substudy 2). For exploratory purposes, the study will examine effects on additional measures of cognition, functioning and self-ratings scales (tertiary outcomes).

The investigators will compare the combination of altitude-like hypoxia (12%) and cognitive training with (1) hypoxia with no training, (2) cognitive training under normal oxygen levels (normoxia; 20%), and (3) normoxia with no training in healthy individuals (substudy 1). For patients with mood disorders (substudy 2) the effects of altitude-like hypoxia (12%) and cognitive training are compared to treatment as usual (TAU).

DETAILED DESCRIPTION:
ALTIBRAIN aims to test a novel model, linking altitude-like oxygen manipulations, endogenous erythropoietin (EPO) in the brain, neuroplasticity and cognition. Specifically, ALTIBRAIN will determine whether upregulation of endogenous brain EPO by altitude-like hypoxia cognition training is a fundamental mechanism of enduring neuroplasticity and long-lasting cognitive improvement in humans. This will be investigated in healthy individuals (substudy 1) and symptomatically stable patients with mood disorders (depression or bipolar disorder; substudy 2).

Substudy 1 involves four intervention groups: (1) altitude-like hypoxia (12%) combined with cognitive training, (2) hypoxia with no training, (3) cognitive training under normoxia (20%), and (4) normoxia with no training. Participants are randomised in blocks of four and undergo interventions in these groups for practical reasons. During the 3-weeks treatment, participants breathe 12% ambient oxygen (≈4400 meters altitude) or normal sea-level oxygen (20%) in a treatment room, 3.5 hours daily, six days per week. On iPads, they perform cognitive training or matched control games without cognitive benefits. Cognitive training is interleaved by short breaks, during which the participants can relax or walk on a treadmill inside the room. Participants undergo cognition assessments in weeks 1 (baseline), 4 and 8 and functional and structural MRI in weeks 1 and 8, when red blood cells are comparable between groups. A subgroup will also undergo PET scanning in week 4.

In substudy 2, patients are randomized to either (1) altitude-like hypoxia (12%) combined with cognitive training, 3.5 hours daily, five-six days per week for three weeks or (2) treatment as usual (TAU). After completed testing, patients in the TAU group undergo the 3-week active intervention, followed by an additional session of neurocognitive testing in the week after treatment completion. All remaining study procedures are identical to substudy 1.

The power calculation was based on the primary hypothesis that altitude-like hypoxia combined with cognitive training produces robust sustained cognitive improvement compared with normoxia and no training. To accommodate for up to a 15% drop-out, we will include 30 participants per group; i.e., 120 healthy individuals and 60 patients to obtain complete data for minimum 26 participants per group, i.e., 104 healthy individuals and 52 patients.

ELIGIBILITY:
Inclusion Criteria (substudy 1):

* 18-50 years
* No psychiatric history
* Fluency in Danish

Inclusion Criteria (substudy 2):

* 18-65 years
* International Classification of Diseases (ICD)-10 diagnosis of Bipolar Disorder or depression confirmed with the Schedules for Clinical Assessment in Neuropsychiatry (SCAN)
* Fluency in Danish
* Partial or full remission (defined as a score of ≤14 on the Hamilton Depression Rating Scale 17-items (HDRS-17) and the Young Mania Rating Scale (YMRS)
* Objectively-verified cognitive impairment according to Screen for Cognitive Impairment in Psychiatry (SCIP) and/or self-reported cognitive impairment measured with Cognitive Complaints in Bipolar disorder Rating Assessment (COBRA). For SCIP, their performance must be ≥0.5 standard deviations (SD) below their demographically adjusted expected total SCIP score or on minimum 2 SCIP subtest scores. For COBRA, patients must report substantial cognitive impairment defined as a score ≥14.

Common Exclusion Criteria:

* Schizophrenia or schizoaffective disorder
* Neurological disorder
* Alcohol or substance abuse
* History of serious head trauma
* Previous altitude sickness
* Heart disease
* Diabetes
* Renal failure
* Untreated/insufficiently treated hypertension
* Thromboses or thromboembolic events
* First-degree family with thromboembolic events before age 60
* Pregnancy
* Breastfeeding
* Smoking or use other nicotine products regularly
* BMI>30
* Electroconvulsive therapy (ECT) 3 months prior to participation
* Dyslexia
* Claustrophobia (MRI scans)
* Pacemaker and/or other MRI incompatible metal implants (MRI scans)
* Participation in experiments with radioactivity (>10 mSv) within the last year (PET scans)
* Significant occupational exposure to radioactivity (PET scans)
* Medication incompatible with study aims (e.g., SV2A binding agents; PET scans)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Cognitive composite score | Baseline, week 4 (end of treatment. Primary outcome assessement time point), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  A cognitive composite based on an average of Z-transformed scores from the Rey Auditory Verbal Learning Test (RAVLT), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding, verbal fluency with the letter "D", WAIS-III Letter-Number Sequencing, Trail Making Test B (TMT B) and Rapid Visual Information Processing (RVP) speed for correct responses from Cambridge Cognition (CANTAB). No score range. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
"Mean choices to correct" in One Touch Stockings of Cambridge (OTS) from Cambridge Cognition (CANTAB) | Baseline, week 4 (end of treatment. Secondary outcome assessement time point), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing executive functions. No score range. Lower scores mean a better outcome.
Dorsal prefrontal cortex activity during spatial N-back | Baseline, week 8
  Functional magnetic resonance imaging (fMRI) measure of brain activity during a working memory task.
ONLY IN PATIENTS (SUBSTUDY 2): Cognition Assessement in Virtual Reality (CAVIR) test: Composite score | Baseline, week 8 (secondary outcome assessment time point) (+end of treatment follow-up for patients in treatment as usual group)
  Self-administered 360º immersive virtual reality test in a kitchen, where the participant's abilities to plan and prepare a meal are assessed. The test involves five subtasks probing verbal memory, executive functions, processing speed, working memory and sustained attention, which are summarized in a composite score. No score range. Higher scores mean a better outcome.

OTHER OUTCOMES:
Rey Auditory Verbal Learning Test | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing verbal memory. Outcomes include total recall (score range 0-75), immediate recall (score range 0-15), and delayed recall (score range 0-15). Higher scores mean a better outcome
Trail Making Test Part A | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing attention and processing speed. Scored as time to complete. A higher time means a worse outcome.
Trail Making Test Part B | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing executive functions. Scored as time to complete. A higher time means a worse outcome.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing attention. Score range 0-89. Higher scores mean a better outcome.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Digit Span | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing executive functions. Score range 0-16. Higher scores mean a better outcome.
Wechsler Adult Intelligence Scale (WAIS)-III Letter-Number Sequencing | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing executive functions. Score range 0-21. Higher scores mean a better outcome.
Verbal fluency with the letter "D" and 'S" | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing executive functions. No score range. Higher scores mean a better outcome.
Rapid Visual Information Processing (RVP) from Cambridge Cognition (CANTAB) | Baseline, week 4 (end of treatment) and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing sustained attention. Outcomes include signal detection (score range 0-1, higher scores mean a better outcome), probability of hit (score range 0-1, higher scores mean a better outcome), total false alarms (score range 0-546, higher scores mean a worse outcome), and latency to correct (score range 100-1900, higher scores mean a worse outcome).
Spatial Working Memory (SWM) from Cambridge Cognition (CANTAB) | Baseline, week 4 (end of treatment) and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing visual working memory. Outcomes include errors (score range 0-153, higher scores mean a worse outcome) and strategy (score range 3-26, higher scores mean a worse outcome).
One Touch Stockings of Cambridge (OTS) from Cambridge Cognition (CANTAB) | Baseline, week 4 (end of treatment) and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing executive functions. Apart from mean choices to correct (secondary outcome), outcomes include problems solved on first choice (score range 1-15, higher scores mean a better outcome), and latency to correct (no score range, higher scores mean a worse outcome).
Emotion Recognition Task (ERT) from Cambridge Cognition (CANTAB) | Baseline, week 4 (end of treatment) and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing social cognition. Outcomes include reaction time (no score range, higher scores mean a worse outcome) and hit rate (score range 0-1, higher scores mean a better outcome).
Wisconsin Card Sorting Task (WCST) | Baseline, week 4 (end of treatment) and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Neuropsychological test assessing executive function. No score range. Higher scores mean a worse outcome.
Cognition Assessement in Virtual Reality (CAVIR) test | Baseline and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  The CAVIR test is a self-administered 360º immersive VR test in a kitchen, where the participant's abilities to plan and prepare a meal are assessed. The test involves five subtasks probing verbal memory, executive functions, processing speed, working memory and sustained attention. No score range. Higher scores mean a better outcome.
The Assessment of Quality of Life (AQoL) | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Questionnaire on quality of life. Score range 33-176. Higher scores mean a worse outcome.
World Health Organization Quality of Life (WHOQoL-BREF) | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Questionnaire on quality of life. Score range 26-130. Higher scores mean a better outcome.
Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA) | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Questionnaire on subjective cognitive complaints. Score range 0-48. Higher scores mean a worse outcome.
Work and Social Adjustment Scale (WSAS) | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Questionnaire on occupational functioning. Score range 0-40. Higher scores mean a worse outcome.
Sheehan Disability Scale (SDS) | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Questionnaire on daily functioning. Score range 0-30. Higher scores mean a worse outcome.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 4 (end of treatment), and week 8 (+end of treatment follow-up for patients in treatment as usual group)
  Questionnaire on sleep quality. Score range 0-21. Higher scores mean a worse outcome.
ONLY IN PATIENTS (SUBSTUDY 2): Functional Assessment Short Test (FAST) | Baseline and week 8
  Clinical interview on daily functioning. Score range 0-72. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla W Miskowiak, DMSc, DPhil, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Neurocognition and Emotion in Affective Disorders (NEAD) Centre, University of Copenhagen and Psychiatric Centre Copenhagen, Frederiksberg hospital, Copenhagen, Capital Region of Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miskowiak KW, Damgaard V, Schandorff JM, Macoveanu J, Knudsen GM, Johansen A, Plaven-Sigray P, Svarer C, Fussing CB, Cramer K, Jorgensen MB, Kessing LV, Ehrenreich H. Effects of cognitive training under hypoxia on cognitive proficiency and neuroplasticity in remitted patients with mood disorders and healthy individuals: ALTIBRAIN study protocol for a randomized controlled trial. Trials. 2024 Oct 3;25(1):648. doi: 10.1186/s13063-024-08463-5. PMID 39363230